CLINICAL TRIAL: NCT01545154
Title: Phase II Study of The Use of Transperineal Ultrasound for Radiation Therapy Treatment Planning and Image Guidance in the Treatment of Prostate Cancer
Brief Title: The Use of Transperineal Ultrasound for Radiation Therapy Treatment Planning and Image Guidance in the Treatment of Prostate Cancer
Status: Completed | Type: Observational
Sponsor: H. James Wallace, MD (Other)
Collaborators: Elekta Limited (Industry)
Responsible Party: Sponsor-Investigator, H. James Wallace, MD, Principal Investigator, University of Vermont Medical Center
Organization: University of Vermont Medical Center (Other)
Other Study IDs: CHRMS M12-073
Record Dates: First submitted 2012-02-29; First posted 2012-03-06 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Prostate Cancer
  Interventions: Device: Transperineal Ultrasound

INTERVENTIONS:
Device: Transperineal Ultrasound

SUMMARY:
This study is being done to find out if transperineal ultrasound (TPUS) can help define the prostate gland for radiation treatment planning and improve upon current methods of image guidance for the treatment of prostate cancer. For the patient, TPUS involves the placement of an ultrasound probe on the perineum, the skin between the scrotum and anus, while they are lying on their back in the position they will receive their treatment. Image-guidance is required for the treatment of prostate cancer because the prostate shifts position depending on how full the bladder and rectum are. Image-guided radiation therapy has been done at Fletcher Allen Health Care for approximately three years. Most commonly, transabdominal ultrasound images are obtained every day and compared to an ultrasound that was done on the day of treatment planning. Adjustments in radiation field position can be done on a daily basis by comparing these images. Transperineal ultrasound has never been used for image-guidance. The investigators completed an earlier study and have developed a TPUS device and process that allow us to get clear ultrasound pictures of the prostate gland. The TPUS has three potential advantages over the transabdominal method the investigators currently use:

1. Transabdominal ultrasound can be a challenge for some men. A full bladder helps us get clearer images, however it is difficult for some men with prostate cancer to comfortably keep a full bladder. It is also particularly difficult to get good images in larger men who have long distances from the skin surface to the prostate gland. TPUS is not dependent on a man having a full bladder and should be less dependent on the size of the man.
2. TPUS images and the planning CT images can be acquired simultaneously. This is not possible with the abdominal probe because it gets in the way of the CT machine. Simultaneous imaging eliminates the possibility of the prostate gland shifting positions during the time between imaging studies.
3. TPUS can be in place and acquire images during patient treatment (the abdominal probe gets in the way of the treatment machine) and may in the future allow us to watch the prostate gland during treatment. If the investigators discover that they can accurately view the prostate gland in real time, TPUS may ultimately allow us to treat even smaller radiation fields and possibly decrease the risk of radiation complications.

Patients in this study will be treated for their prostate cancer with the standard image guidance techniques used at Fletcher Allen Health Care: transabdominal ultrasound and/or X-ray imaging of gold marker seeds that have been placed the prostate gland. In addition to standard care, all men in this study will have TPUS and CT scans done a total of four times over 12 weeks to compare these methods of prostate localization over the course of radiation treatments. Some men may choose to take part in an additional study that will also include MRI of the pelvis to compare with the TPUS and CT. Because the prostate gland can be more clearly defined on MRI, some institutions (not Fletcher Allen) routinely have patients with prostate cancer get MRI scans for treatment planning. This has not been proven to improve the care of men with prostate cancer and it is possible that TPUS will provide similarly clear images. The potential advantages to TPUS imaging for prostate localization over MRI include the fact that it is done at the same time as the CT for treatment planning (so eliminates the possibility of movement of the prostate gland from the time of the MRI to the time of the CT) and can be done at a much lower cost.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of prostate cancer

Exclusion Criteria:

* Prostatectomy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males with prostate cancer, 18+
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2012-02; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Fletcher Allen Health Care, Burlington, Vermont, United States